CLINICAL TRIAL: NCT04259268
Title: Evaluation of the Quality of Preoperative Information Obtained Through Preanestes@s, a Web Based Application: Paired Comparison of a Web Based Questionnaire, a Virtual Non Face to Face Assessment and Outpatient Visit
Brief Title: Evaluation of the Quality of Preoperative Information Obtained Through Preanestes@s, a Web Based Application
Acronym: Preanestes@s
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: PIN-0224-2018
Record Dates: First submitted 2020-01-02; First posted 2020-02-06 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Mobile Applications; Internet-Based Intervention; Preoperative Period
Keywords: Patient Health Questionnaire; Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Web based questionnaire: Information registered by patient in the web based questionnaire
  Interventions: Other: Quality of preoperative information register
- Outpatient assessment: Information registered by the anesthesiologist and based on the web based questionnaire, the electronic records of patient and the "face to face" interview
  Interventions: Other: Quality of preoperative information register; Other: Suitability of information contained in the informed consent
- Virtual assessment: Information registered by the anesthesiologist and based on the web based questionnaire and the electronic records of patient
  Interventions: Other: Quality of preoperative information register; Other: Suitability of information contained in the informed consent

INTERVENTIONS:
Other: Quality of preoperative information register — Register of principal (grade ASA classification) and secondary variables (allergies, antiplatelet or blood thinners prescriptions, cardiovascular diseases, present medication)
Other: Suitability of information contained in the informed consent — Register of information regarding specific individual risks and personal data (patient and doctor identification and signature)
  Groups: Outpatient assessment; Virtual assessment

SUMMARY:
In this prospective and paired study, the investigators evaluate whether the preoperative information recorded through a web based questionnaire together with a virtual non face to face patient assessment based on the information recorded by the questionnaire and the electronic records of patients is of a comparable quality to that obtained with the traditional outpatient interview.

DETAILED DESCRIPTION:
Preanestes@s is a web based application conceived to lead patients through the preoperative period. The application includes a patient interface which offers general and individualized information on the perioperative process, with the possibility of generating a dynamic interaction between patients and medical staff. Patient interface incorporates a web based preoperative questionnaire that once fully completed, will automatically indicate which preoperative tests are necessary and will address patients to a virtual (non face to face) consultation or to traditional outpatient assessment. Both virtual and outpatient assessment will be performed by an anesthesiologist. The web based questionnaire will automatically assign patients an ASA grade (from the American Society of Anesthesia Physical Status Classification); this being the determining variable, although not the only one, when directing patients to the virtual or face-to-face consultation.The questionnaire therefore serves both for collection of clinical information, and as a patient classification tool as well.

Virtual assessment will be the performed by evaluating both the filled web based questionnaire together with participants´ electronic records. Face to face assessment will be performed in the traditional way by means of an interview with the participant together with the consultation of participant´s previous electronic records.

The virtual assessment will be reserved for participants without significant comorbidity, which would correspond to patients classified as grade ASA 1-2; this means participants without diseases or with diseases that do not significantly compromise the integrity of the participant: well-controlled hypertension, active smoking without major lung disease, non-morbid obesity, etcetera. Participants with significant comorbidity (grade ASA ≥ 3), will always be referred to a face-to-face consultation.

This study has been approved by the local Ethics Committee -Comité de Ética e Investigación de Huelva-and signed by its Secretary María Dolores Santos Rubio, date 18.12.2019.

The investigators´objective is to evaluate whether the information recorded through the web based questionnaire and the virtual assessment is of a comparable quality to that obtained with the gold standard, the traditional face to face outpatient interview.To answer this question, the investigators have designed a prospective paired stud. After obtaining the correspondent informed consent, the investigators will ask participants to fill the web based questionnaire. In participants submitted to virtual assessment after completing the questionnaire, an investigator will perform the virtual preoperative evaluation; these participants will also be submitted to traditional outpatient evaluation in order to compare both types of evaluation. In participants submitted to outpatient assessment, the investigators will compare traditional face to face visit with the questionnaire information.

The investigators will study the degree of concordance in the recording of preoperative variables between different methods (web based questionnaire, virtual assessment and outpatient assessment). The variables to be analysed are described in the Outcomes Measure section.

The investigators will also compare the suitability of information recorded in the anesthetic paper based informed consent (pIC) versus the electronic informed consent (eIC) included in the application. The investigators hypothesis is that Preanestes@s web based questionnaire together with the virtual assessment allows a collection of preoperative information at least as reliable as the classic face to face interview format.

Statistical analysis: the investigators will analyze the agreement between observers (Interrater reliability) for the qualitative variables selected, making comparisons between the different methods of recording information for each variable included in the analysis (study of paired samples). The investigators will use the Fleiss Kappa coefficient to study the concordance in the measurement of the categorical variables.

For the estimation of the sample size, the investigators will group the categories ASA grade 1-2 versus ASA grade 3 and 4, since in the model proposed , the ASA grade ≥ 3 leads patients to a face-to-face outpatient visit. The investigators assume, therefore, the ASA grade as a dichotomous variable (ASA ≥ 3 present or absent). With these considerations, and based on the Table of Concordance of the work of Sankar et al and their results (Kappa index 0.68 (95% CI 0.67-0.69)), the investigators estimate a sample size of 318 patients for a Kappa index of 0.68 with a precision level of 0.08 and an 95% CI. The investigators will recruit, in principle, a total of 382 participants, assuming a potential loss of 20% of the patients initially included.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients submitted to programmed interventions under anesthetic care in Hospital Universitario Virgen del Rocío

Exclusion Criteria:

* Patients unable to fully understand the informed consent
* Urgent or emergent surgery
* Patients submitted to cataract surgery, as far as this procedure is attended by specific clinical pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients submitted to programmed interventions under anesthetic care in Hospital Universitario Virgen del Rocío
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Change in ASA grade classification | 60 days before intervention (web-based questionnaire) and 30 days before intervention (virtual and outpatient assessment)
  Comparison of the ASA grade assigned automatically when patients fill the web based questionnaire versus that assigned by the anesthesiologist following the virtual or outpatient assessment

SECONDARY OUTCOMES:
Change in the register of any allergies | 60 days before intervention (web-based questionnaire) and 30 days before intervention (virtual and outpatient assessment)
  Comparison of the presence of any allergies registered by patient in the web based questionnaire those included in patient´s electronic records or registered by the anesthesiologist following the virtual or outpatient assessment
Change in the register of antiplatelet or blood thinners | 60 days before intervention (web-based questionnaire) and 30 days before intervention (virtual and outpatient assessment)
  Comparison in the register of antiplatelet or blood thinners either by patient through the web based questionnaire versus those registered in patient´s electronic records or by the anesthesiologist following the virtual or outpatient assessment
Change in the register of cardiovascular diseases | 60 days before intervention (web-based questionnaire) and 30 days before intervention (virtual and outpatient assessment)
  Comparison in the register of cardiovascular diseases registered either by patient through the web based questionnaire or by the anesthesiologist following the virtual or outpatient assessment
Register of the ASA grade in the informed consent form | The day of intervention
  Comparison in the register of the ASA grade either in the paper based informed consent versus the electronic informed consent
Register of personal name and surname in the informed consent form | The day of intervention
  Comparison in the register of the names and surnames of both patient and anesthesiologist either in the paper based informed consent versus the electronic informed consent

CONTACTS AND LOCATIONS:
Overall Officials: Manuel de la Matta, MD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Hert S, Staender S, Fritsch G, Hinkelbein J, Afshari A, Bettelli G, Bock M, Chew MS, Coburn M, De Robertis E, Drinhaus H, Feldheiser A, Geldner G, Lahner D, Macas A, Neuhaus C, Rauch S, Santos-Ampuero MA, Solca M, Tanha N, Traskaite V, Wagner G, Wappler F. Pre-operative evaluation of adults undergoing elective noncardiac surgery: Updated guideline from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2018 Jun;35(6):407-465. doi: 10.1097/EJA.0000000000000817. PMID 29708905
- [Background] Katz RI, Dexter F, Rosenfeld K, Wolfe L, Redmond V, Agarwal D, Salik I, Goldsteen K, Goodman M, Glass PS. Survey study of anesthesiologists' and surgeons' ordering of unnecessary preoperative laboratory tests. Anesth Analg. 2011 Jan;112(1):207-12. doi: 10.1213/ANE.0b013e31820034f0. Epub 2010 Nov 16. PMID 21081771
- [Background] Zaballos M, Lopez-Alvarez S, Argente P, Lopez A; Grupo de Trabajo de Pruebas Preoperatorias. Preoperative tests recommendations in adult patients for ambulatory surgery. Rev Esp Anestesiol Reanim. 2015 Jan;62(1):29-41. doi: 10.1016/j.redar.2014.07.007. Epub 2014 Aug 18. English, Spanish. PMID 25146773
- [Background] Arias A, Benitez S, Canosa D, Borbolla D, Staccia G, Plazzotta F, Casais M, Michelangelo H, Luna D, Bernaldo de Quiros FG. Computerization of a preanesthetic evaluation and user satisfaction evaluation. Stud Health Technol Inform. 2010;160(Pt 2):1197-201. PMID 20841873
- [Background] Applegate RL 2nd, Gildea B, Patchin R, Rook JL, Wolford B, Nyirady J, Dawes TA, Faltys J, Ramsingh DS, Stier G. Telemedicine pre-anesthesia evaluation: a randomized pilot trial. Telemed J E Health. 2013 Mar;19(3):211-6. doi: 10.1089/tmj.2012.0132. Epub 2013 Feb 5. PMID 23384334
- [Background] Blanco Vargas D, Faura Messa A, Izquierdo Tugas E, Santa-Olalla Bergua M, Noguera Sopena MM, Manoso Noriego M. [Online versus non-standard face to face preoperative assessment: cost effectiveness]. Rev Esp Anestesiol Reanim. 2012 Aug-Sep;59(7):350-6. doi: 10.1016/j.redar.2012.05.039. Epub 2012 Jul 10. Spanish. PMID 22784647
- [Background] de la Matta Martin M, Forastero Rodriguez A, Lopez Romero JL. [Evaluation of a new computerized recording system for preoperative assessment data]. Rev Esp Anestesiol Reanim. 2011 Oct;58(8):485-92. doi: 10.1016/s0034-9356(11)70123-2. Spanish. PMID 22141216
- [Background] Ludbrook G, Seglenieks R, Osborn S, Grant C. A call centre and extended checklist for pre-screening elective surgical patients - a pilot study. BMC Anesthesiol. 2015 May 19;15:77. doi: 10.1186/s12871-015-0057-1. PMID 25985775
- [Background] Law TT, Suen DT, Tam YF, Cho SY, Chung HP, Kwong A, Yuen WK. Telephone pre-anaesthesia assessment for ambulatory breast surgery. Hong Kong Med J. 2009 Jun;15(3):179-82. PMID 19494372
- [Background] Lozada MJ, Nguyen JT, Abouleish A, Prough D, Przkora R. Patient preference for the pre-anesthesia evaluation: Telephone versus in-office assessment. J Clin Anesth. 2016 Jun;31:145-8. doi: 10.1016/j.jclinane.2015.12.040. Epub 2016 Apr 15. PMID 27185698
- [Background] Goodhart IM, Andrzejowski JC, Jones GL, Berthoud M, Dennis A, Mills GH, Radley SC. Patient-completed, preoperative web-based anaesthetic assessment questionnaire (electronic Personal Assessment Questionnaire PreOperative): Development and validation. Eur J Anaesthesiol. 2017 Apr;34(4):221-228. doi: 10.1097/EJA.0000000000000545. PMID 27798453
- [Background] Sankar A, Johnson SR, Beattie WS, Tait G, Wijeysundera DN. Reliability of the American Society of Anesthesiologists physical status scale in clinical practice. Br J Anaesth. 2014 Sep;113(3):424-32. doi: 10.1093/bja/aeu100. Epub 2014 Apr 11. PMID 24727705
- [Background] ASA House of Delegates/Executive Committee. ASA Satandards and Guidelines. ASA Physical Status Classification System.2014. https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
- [Background] Kinley H, Czoski-Murray C, George S, McCabe C, Primrose J, Reilly C, Wood R, Nicolson P, Healy C, Read S, Norman J, Janke E, Alhameed H, Fernandes N, Thomas E. Effectiveness of appropriately trained nurses in preoperative assessment: randomised controlled equivalence/non-inferiority trial. BMJ. 2002 Dec 7;325(7376):1323. doi: 10.1136/bmj.325.7376.1323. PMID 12468478
- [Derived] de la Matta M, Alonso-Gonzalez M, Moreno-Conde J, Salas-Fernandez S, Lopez-Romero JL; Preanestesas study investigators. Development and patient acceptance of Preanestes@s, a web-based application and electronic questionnaire for preoperative assessment. A prospective cohort study. Rev Esp Anestesiol Reanim (Engl Ed). 2022 Aug-Sep;69(7):383-392. doi: 10.1016/j.redare.2022.01.002. Epub 2022 Jul 20. PMID 35871145